CLINICAL TRIAL: NCT00032786
Title: A Phase 3, International, Multicenter, Double-blind, Placebo-controlled Study of the Efficacy, Safety, and Tolerability of Intravenous Antegren (Natalizumab) in Maintaining Clinical Response and Remission in Subjects With Crohn's Disease
Brief Title: Safety and Efficacy of Natalizumab in the Treatment of Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CD303
Record Dates: First submitted 2002-04-03; First posted 2002-04-04 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2012-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Natalizumab

INTERVENTIONS:
Drug: natalizumab

SUMMARY:
The purpose of this study is to determine the safety and efficacy of natalizumab in individuals diagnosed with moderate to severely active Crohn's disease. It is thought that natalizumab may stop the movement of certain cells, known as white blood cells, into bowel tissue. These cells are thought to cause damage in the bowel leading to the symptoms of Crohn's disease.

ELIGIBILITY:
Male and female patients at least 18 years of age who have at least a six-month history of Crohn's disease and who are currently experiencing moderate to severely active Crohn's disease. Women must not be breastfeeding or pregnant, and must not become pregnant during this study. Patient enrollment requires previous participation in study AN100226-CD301 (please refer to the clinical trial listing for CD301).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-03; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

REFERENCES:
- [Result] Sandborn WJ, Colombel JF, Enns R, Feagan BG, Hanauer SB, Lawrance IC, Panaccione R, Sanders M, Schreiber S, Targan S, van Deventer S, Goldblum R, Despain D, Hogge GS, Rutgeerts P; International Efficacy of Natalizumab as Active Crohn's Therapy (ENACT-1) Trial Group; Evaluation of Natalizumab as Continuous Therapy (ENACT-2) Trial Group. Natalizumab induction and maintenance therapy for Crohn's disease. N Engl J Med. 2005 Nov 3;353(18):1912-25. doi: 10.1056/NEJMoa043335. PMID 16267322